CLINICAL TRIAL: NCT00688246
Title: The Influence of Five Years of Exemestane on Bone Mineral Density in Postmenopausal Women at Increased Risk of Developing Breast Cancer
Brief Title: Bone Mineral Density in Postmenopausal Women at Increased Risk of Breast Cancer And Who Are Receiving Exemestane on MAP3
Status: Completed | Type: Observational
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Other Study IDs: MAP3B; CAN-NCIC-MAP3B (Registry Identifier: NCI US - Physician Data Query); PFIZER-NCIC-MAP3B (Other: Pfizer); CDR0000586285 (Other: PDQ)
Record Dates: First submitted 2008-05-30; First posted 2008-06-02 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biologic sample preservation procedure — Increased bone turnover may be a risk factor for fracture [Lønning 2005]. However, it is uncertain whether markers of bone resorption and markers of bone formation are both associated with fracture risk [Looker 2000]. Therefore, we will measure bone formation and bone resorption markers at baseline, year 1 and year 5. Blood specimens will be shipped to and stored in a central laboratory for future assays of bone biomarkers. For markers of bone formation, the N-terminal Propeptide of Type I Collagen (PINP) will be measured. For bone resorption markers, serum levels of cross-linked N-telopeptides of type I collagen (NTx) will be measured. Note: Subjects must fast 12-14 hours prior to blood draw.
Procedure: dual x-ray absorptometry — BMD of the spine (L1-L4) and total hip will be done within 12 months prior to randomization to the MAP.3 core protocol. BMD by DEXA of the spine (L1-L4) and total hip will be repeated at year 2 and year 5 of the MAP.3 core study on the same Lunar or Hologic scanner.

SUMMARY:
RATIONALE: Learning about the effect of exemestane on bone mineral density in postmenopausal women at increased risk of breast cancer may help plan treatment, decrease the risk of broken bones, and help patients live more comfortably.

PURPOSE: This research study is measuring bone mineral density in postmenopausal women at increased risk of developing breast cancer who are receiving exemestane on clinical trial CAN-NCIC-MAP3.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the percentage change in bone mineral density (BMD) as measured by dual x-ray absorptometry (DEXA) scans of the spine (L1-L4) and total hip 2 years after randomization (and registration to the MAP.3B protocol).

Secondary

* To assess the percentage change in BMD as measured by DEXA scans of the spine (L1-L4), and total hip 5 years after randomization (and registration to the MAP.3B protocol).
* To compare the proportion of women who develop BMD of the spine (L1-L4) and total hip below the absolute threshold value for osteoporosis (T score ≤ -2.5 SD below the mean peak bone mass in young women) in the treatment groups.
* To examine the pattern of changes in BMD parameters and bone biomarkers (i.e., PINP and NTx) over time and the impact of covariants using exploratory longitudinal analyses.
* To compare the proportion of women who develop clinical skeletal fractures in the treatment groups.

OUTLINE: Patients undergo bone mineral density (BMD) measurement by dual x-ray absorptometry (DEXA). Blood specimens are collected at baseline and at 1 year, and 5 years and stored in a central laboratory for future assays of the bone biomarkers.

If the subject withdraws from the core MAP.3 study before 5 years, a bone density measurement and serum for bone biomarkers is obtained unless performed within the past 3 months. Patients may continue to be followed on the MAP.3 core study for fractures (and other MAP.3 study endpoints) for a minimum of 5 years after randomization.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk of developing breast cancer and enrolled on clinical trial CAN-NCIC-MAP3
* Bone mineral density (BMD) (as measured by dual x-ray absorptometry [DEXA] scans within 12 months prior to randomization to the core protocol [MAP.3]) T score > -2.0 standard deviation (i.e., 2.0 standard deviations below the average peak BMD of a young adult woman) of spine (L1-L4) and total hip
* Serum for bone biomarkers (i.e., serum N-telopeptide and serum amino-terminal procollagen 1 extension peptide) must have been obtained within 8 weeks prior to registration to the study

PATIENT CHARACTERISTICS:

* Postmenopausal, defined as one of the following:

  * Over 50 years of age with no spontaneous menses for at least 12 months before study entry
  * 50 years of age or under with no menses (spontaneous or secondary to hysterectomy) for at least 12 months before study entry AND with follicle-stimulating hormone level within postmenopausal range
  * Underwent prior bilateral oophorectomy
* Available for collection of serum samples and BMD (DEXA) scans at the protocol defined times (i.e., have BMD scans at years 2 and 5 at the same site)
* No history of fragility fractures (i.e., a broken bone that occurs with a fall from a standing height or lesser amount of trauma)
* No malabsorption syndrome (e.g., untreated celiac disease, clinically relevant vitamin D deficiency, or active hyper- or hypoparathyroidism)
* No Paget disease or other metabolic bone diseases (e.g., osteomalacia or osteogenesis imperfecta)
* No Cushing disease or other pituitary diseases
* No inflammatory disease(s) (e.g., inflammatory bowel disease, rheumatoid arthritis, lupus, psoriasic arthritis, ankylosing spondylitis, or autoimmune hepatitis)

PRIOR CONCURRENT THERAPY:

* More than 3 months since prior bone drugs, such as bisphosphonates, teriparatide (parathyroid hormone [PTH]), sodium fluoride, calcitonin (Miacalcin®), strontium, or high-dose vitamin D (i.e., vitamin D3 > 2,000 IU/day or calcitriol)
* No prior bisphosphonate therapy duration of more than 6 months total during lifetime
* No concurrent anabolic or chronic oral corticosteroids (the equivalent of 5 mg of prednisone a day or higher for more than 2 weeks within the past 6 months and will likely require ongoing therapy)
* Concurrent inhaled steroids allowed
* No concurrent medication that may have an effect on study endpoints for this study, including any of the following:

  * Anticonvulsants
  * Sodium fluoride at daily doses > 5 mg/day for a period exceeding 1 month
  * Anabolic steroids
  * Teriparatide (parathyroid hormone)
  * Bisphosphonates, except for women who develop osteoporosis while on this study; these patients may be advised to start bone medication (i.e., strontium, calcitonin, or high-dose Vitamin D (i.e., Vitamin D3 > 2000 IU/day or calcitriol) at the discretion of their physician

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible women consenting to be randomized to the core MAP.3 trial will be approached for participation in this companion study. They must have an acceptable quality BMD scan by DEXA taken within 12 months prior to randomization to MAP.3. A BMD T-score > -2.0 SD (i.e. 2.0 standard deviations below the average peak BMD of a young adult woman) has been established as the study population cut-off because postmenopausal women who have BMD T-scores as low as or lower than - 2.0 SD are currently recommended to consider pharmacological therapies for their bones
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2008-07-10 (Actual); Primary Completion 2011-10-31 (Actual); Study Completion 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density (BMD) as measured by dual x-ray absorptometry (DEXA) scans of the spine (L1-L4) and total hip 2 years after randomization | 2 years

SECONDARY OUTCOMES:
Change in BMD as measured by DEXA scans of the spine (L1-L4) and total hip 5 years after randomization on CAN-NCIC-MAP3 | 5 years
Changes in markers of bone formation and resorption 1 and 5 years after randomization on CAN-NCIC-MAP3 | 5 years
Development of osteoporosis either by sustaining a fragility fracture or by having a BMD T-score at or lower than - 2.5 SD at the spine (L1-L4) or total hip | 2 years
Number of clinical skeletal fractures by radiology report | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (18):
- United States (13):
  - Los Angeles Biomedical Research Institute, Torrance, California
  - The George Washington University, Washington D.C., District of Columbia
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Suburban Hospital Cancer Program, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hutzel Women's Health Specialists, Detroit, Michigan
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - University of Oklahoma, Oklahoma City, Oklahoma
  - The Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Fletcher Allen Health Care, Burlington, Vermont
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Univ. of Wisconsin Center for Women's Health and, Madison, Wisconsin
- Canada (5):
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No